CLINICAL TRIAL: NCT01967966
Title: A PHASE 1 STUDY TO INVESTIGATE THE ABSOLUTE BIOAVAILABILITY OF GDC-0032 AND THE ABSORPTION, METABOLISM, AND EXCRETION OF [14C]-GDC-0032 IN HEALTHY MALE SUBJECTS
Brief Title: A Bioavailability and Pharmacokinetic Study of GDC-0032 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP28755
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

ARMS (2):
- Bioavailability (Experimental)
  Interventions: Drug: GDC-0032
- Elimination & PK (Experimental)
  Interventions: Drug: GDC-0032

INTERVENTIONS:
Drug: GDC-0032 — Single oral dose
Drug: GDC-0032 — Single IV dose
  Arms: Bioavailability

SUMMARY:
This 2-arm, open-label, non-randomized study will investigate the absolute bioavailability, pharmacokinetics, mass balance, and routes of elimination of GDC-0032 as well as its safety in healthy volunteers. Patients will receive either a single oral dose of GDC-0032 followed by a 14C-labeled IV dose of GDC-0032 or a single oral dose of 14C-labelled GDC-0032.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18 to 32 kg/m2, inclusive;
* Healthy, as judged by physician from medical history, 12-lead ECG, vital signs, and clinical laboratory evaluations;
* Agree to use effective contraceptive methods as defined by protocol;
* Negative hepatitis panel and HIV screen;
* Sufficient bowel movements (minimum of 1 per day).

Exclusion Criteria:

* History or clinical manifestation of: any major medical disorders; any food/drug/substance allergies;
* History of stomach or intestinal surgery or resection except for appendectomy and/or hernia repair;
* History of alcoholism or drug addiction within 1 year prior to drug administration;
* Tobacco or nicotine use within 6 months prior to study start;
* Chronic use of gastric acid inhibitors within 6 months of study start or use of gastric acid inhibitors and/or antacids within 1 month prior to drug administration;
* Evidence of malabsorption syndrome or other condition interfering with gastrointestinal absorption;
* Inability or unwillingness to swallow capsules;
* Participation in a drug study in which a drug was administered within 30 days prior to study start;
* Participation in more than one radiolabeled drug study within 12 months preceding drug administration. The previous radiolabeled study drug must have been received more than 6 months prior to this study, and the total exposure from this study and the previous study is less than 5000 mrem whole body annual exposure;
* Exposure to significant radiation within 12 months prior to study start.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability: Absolute bioavailability of GDC-0032 (Area under the concentration-time curve [AUC]) | Days 1 to 11
Elimination & PK: Amount of drug excreted in urine/feces over the sampling interval | Days 1 to 22
Elimination & PK: Maximum concentration (Cmax) of GDC-0032 | Days 1 to 22
Elimination & PK: Area under the concentration-time curve (AUC) | Days 1 to 22
Elimination & PK: Total radioactivity concentrations in whole blood, plasma, urine, and feces. | Days 1 to 22

SECONDARY OUTCOMES:
Elimination & PK: Metabolite identification in plasma, urine, & feces | Days 1 to 22
Safety: Incidence of adverse events | 38 to 49 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Madison, Wisconsin, United States